CLINICAL TRIAL: NCT00696865
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD2624 When Given in Multiple Ascending Oral Doses in Young Healthy Male Japanese Subjects
Brief Title: AZD2624 Multiple Ascending Dose Study in Japan
Acronym: JMAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD, PhD - Medical Science Sr. Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: D0970C00006
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2009-07-16 (Estimated); Status verified 2009-07

CONDITIONS: Healthy; Safety
Keywords: Safety; Tolerability; Phase I
MeSH Terms: interventions — 3-((methylsulfonyl)amino)-2-phenyl-N-(1-phenylpropyl)quinolin-4-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD2624
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2624 — oral suspension, 3 doses
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This multiple ascending dose study will evaluate safety and tolerability after repeated ascending doses of AZD2624

ELIGIBILITY:
Inclusion Criteria:

* Healthy young male Japanese volunteers

Exclusion Criteria:

* Significant illness, as judged by the investigator, within 2 weeks of screening visit or Day 1
* Enrollment in another concurrent investigational study or intake of an investigational drug within 4 months prior to the screening visit or Day 1
* Blood loss in excess of 200 mL within 30 days of screening visit or Day 1, in excess of 400 mL within 90 days of screening visit or Day 1, or in excess of 1200 mL within 1 year of screening visit or Day 1
* Clinically relevant abnormalities in physical examinations, vital signs, clinical chemistry, hematology or urinalysis as judged by the investigator at screening or pre first dose

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-05; Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple ascending oral doses of AZD2624 in young healthy male Japanese subjects compared to placebo by assessment of adverse events, vital signs, physical examinations, laboratory parameters, ECGs and EEGs | All assessments are made at each visit, at least daily, during the study.

SECONDARY OUTCOMES:
To evaluate and characterize the pharmacokinetics of AZD2624 and its metabolites when given orally in multiple ascending doses of AZD2624 to young healthy male Japanese subjects by assessment of drug concentration in plasma | Blood samples will be taken before and after study drug administration.
Identification of genes that influence the disposition, efficacy, safety and tolerability of AZD2624 | A single blood sample will be obtained

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kumagai, MD, PhD, Principal Investigator — Kitasato University East Hospital, Kanagawa, Japan
Locations (1):
- Research Site, Kanagawa, Japan